CLINICAL TRIAL: NCT05473611
Title: Comparison of Open Reduction Internal Fixation and Percutaneous Sacroiliac Screw Fixation in Unstable Posterior Ring Injury of The Pelvic
Brief Title: Open Reduction Internal Versus Percutaneous Sacroiliac Screw Fixation in Unstable Posterior Ring Injury of Pelvic
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Mehmet Koçaslan, Principal investigator, Ataturk University
Other Study IDs: Ataturk University Orthopedic
Record Dates: First submitted 2022-07-22; First posted 2022-07-26 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Orthopedic Disorder
Keywords: instabil pelvic injury, percutaneus sacroiliac screw
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- closed reduction percutaneous fixation method: Patients with closed reduction percutaneous sacroiliac screw fixation of posterior pelvic ring due to unstable pelvic injury
  Interventions: Procedure: closed reduction percutaneous fixation with open reduction internal fixation of the posterior pelvic ring
- open reduction anterior sacroiliac approach: Patients with fixation of the posterior pelvic ring by open reduction anterior approach due to unstable pelvic injury
  Interventions: Procedure: closed reduction percutaneous fixation with open reduction internal fixation of the posterior pelvic ring
- open reduction posterior sacroiliac approach: Patients with fixation of the posterior pelvic ring by open reduction posterior approach due to unstable pelvic injury
  Interventions: Procedure: closed reduction percutaneous fixation with open reduction internal fixation of the posterior pelvic ring

INTERVENTIONS:
Procedure: closed reduction percutaneous fixation with open reduction internal fixation of the posterior pelvic ring — closed reduction percutaneous fixation with open reduction internal fixation of the posterior pelvic ring

SUMMARY:
Surgical trearment of unstable posterior pelvic injuries can be performed with open reduction and internal fixation, closed reduction with percutaneous sacroiliac fixation. Biomechanically, no significant difference was found between the two methods in the literature. The aim of our study is to compare the radiological and clinical functional results of these methods.

DETAILED DESCRIPTION:
Pelvic injuries are usually encountered in patients with polytrauma. These are injuries that need to be treated with a multidisciplinary approach. The primary approach is to stabilize the patient hemodynamically. Mortality rate in pelvic injuries reaches 10-20%.

The pelvis has a ring-shaped structure. It is the sacrum that transfers the load from the lower extremities to the axial spine from this structure. The joint between the sacrum and the ilium, that is, the joint that is exposed to the load, is the sacroiliac joint. For this reason, surgical treatments have been developed to stabilize the posterior pelvic ring, to mobilize the patient as soon as possible, to walk in a balanced way without leg length difference, to prevent loss of work force, and to shorten the hospitalization period. Open reduction internal fixation and closed reduction percutaneous sacroiliac screw fixation surgical methods have been described to ensure the stability of the posterior pelvic ring In this study, we evaluated the radiological and functional results of patients with posterior pelvic ring injuries stabilized by open and closed surgical approaches; We have compiled and summarized the current literature on pelvic injuries. We aimed to contribute to the literature by sharing our knowledge and findings about these difficult, complex and prone surgical techniques.

marks of conformity

1. Surgical intervention for sacroiliac joint fracture-dislocation
2. 18-65 years old patient
3. Patients who come to clinical follow-ups for at least 6 months

ELIGIBILITY:
Inclusion Criteria:

* Surgical intervention for sacroiliac joint fracture-dislocation
* 18-65 years old patient
* Patients who come to clinical follow-ups for at least six months
* not paralyzed

Exclusion Criteria:

* Patients under 18 years of age
* Patients older than 65 years
* Patients who did not come for their follow-up in our clinic
* paralyzed patients
* mentally retarded patients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18-65 years who suffered pelvic injury admitted to Atatürk University Research Hospital
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2022-03-10 (Actual); Primary Completion 2022-11-10 (Estimated); Study Completion 2023-03-12 (Estimated)

PRIMARY OUTCOMES:
functional scoring | at least 6 months
  Grading of outcomes using the clinical functional scoring system for pelvic injuries defined by Majeed
radiological scoring | at least 6 months
  Radiological grading of the treatment process of pelvic fracture with the measurement methods of pelvic plain radiographs defined by Matta and Henderson

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University Faculty of Medicine, Erzurum, Yakutiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided